CLINICAL TRIAL: NCT03556163
Title: Use of Modified Vertical Internal Mattress Suture Versus Simple Loop Interrupted Suture in Modified Widman Flap Surgery- A Randomized Clinical Study.
Brief Title: Modified Vertical Internal Mattress Suture Versus Simple Loop Interrupted Suture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Krishan perio
Record Dates: First submitted 2018-06-02; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Healing Surgical Wounds; Periodontitis
Keywords: Chronic periodontitis; Modified Widman flap surgery; Suturing technique
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Modified vertical internal mattress sutures + MWF surgery.
  Interventions: Procedure: Modified vertical internal mattress sutures + MWF surgery.
- Control Group (Active Comparator): Simple loop interrupted sutures + MWF surgery.
  Interventions: Procedure: Simple loop interrupted sutures + MWF surgery.

INTERVENTIONS:
Procedure: Modified vertical internal mattress sutures + MWF surgery. — Modified vertical internal mattress sutures were given after modified Widman flap surgery.
  Arms: Test Group
Procedure: Simple loop interrupted sutures + MWF surgery. — Simple loop interrupted sutures were given after modified Widman flap surgery.
  Arms: Control Group

SUMMARY:
Aim of study was clinical comparative evaluation of using modified vertical internal mattress suturing technique and simple loop interrupted suturing technique in the outcome of modified Widman flap surgery for the management of chronic periodontitis.

DETAILED DESCRIPTION:
Periodontitis is inflammation of the periodontal tissues resulting in clinical attachment loss, alveolar bone loss, and periodontal pocketing.The destruction of tooth supporting tissues is caused by interaction of bacteria present in the dental plaque and the host .The elimination of bacterial plaque, calculus ,toxic material adhering to tooth surface and other plaque retentive factors can be achieved by nonsurgical and surgical periodontal therapies .The primary objective of periodontal therapy is arresting infection, restoring the lost structure and to maintain healthy periodontium .

The requirement of access for scaling and root planning, pocket depth reduction, correction of gross gingival aberrations ,and establishment of morphology of the dento-gingival area conducive to infection control led to the development of the various surgical procedures. The initial surgical procedures used in periodontal therapy involved excision of the diseased gingival tissue . The main disadvantages of these procedures are unwanted root exposure, poor aesthetics, decrease in width of attached gingiva, excision of frenum attachment and creation of shallow vestibular depth.

Proper management of supracrestal soft tissue flap during suturing appears to be of critical importance in ultimate outcome of surgical periodontal pocket management .A number of studies advocate the proper management of supra-alveolar component of flap in management of infrabony defects employing regenerative techniques with grafts / barrier membrane to minimize postoperative exposure, contamination and/or exfoliation of the grafted material and / or barrier membrane. However review of the available literature does not reveal studies conducted to evaluate the effectiveness of close approximation of flaps by different suturing techniques. Sites with suprabony periodontal pocket depth of 4mm have approximately 6 mm height of unsupported supracrestal soft tissue flap which increases with further increase in pocket depth. Moreover, with advancing probing depth, base of the unsupported soft tissue wall of periodontal pocket comes closer to the musculature in the vestibule, thereby eliciting requirement of a more efficient suturing technique to resist muscle pull for prevention of any disturbance to healing granulation tissue.

The interrupted suturing encompasses two suturing technique; the simple loop and figure of eight. Modified vertical internal mattress suture is a variation of the vertical mattress suture which is especially useful in maximizing wound eversion, reducing dead space, and minimizing tension across the wound. Wound eversion maximize flap approximation. The recommended time for removal of this suture is 5-7 days to reduce the risk of scarring (cross hatching).

Thus the most suitable suturing technique to achieve healing by primary intention and connective tissue reattachment/ periodontal regeneration need to be explored. The present study is intended to determine the influence of the simple interrupted and modified vertical internal mattress suturing technique on the outcome of modified Widman flap surgery .

STUDY DESIGN This randomized clinical interventional study was conducted in Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak.

STUDY POPULATION Out of 172 patients screened from regular OPD in Department of Periodontics and Oral Implantology, the study was conducted in 48 chronic periodontitis participants meeting the eligibility criteria for surgical intervention. 45 patients completed the treatment protocol (28 males and 17 females, mean age: 35.91±7.67 years). Study period was from 01-12-2016 to 31-03-2018.

METHODOLOGY

Periodontal examination

All eligible participants after 8 weeks of phase 1 therapy, were examined in a standardized way using illumination by a standard dental light, a mouth mirror, tweezer, manual calibrated probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA) and explorer. Following parameters were recorded at baseline (day of surgery), after 3 months and 6 months follow up.

* Plaque index (Silness and Loe) (PI)
* Gingival index (Loe and Silness) (GI)
* Bleeding on probing (BOP)
* Probing pocket depth (PPD)
* Clinical attachment level (CAL)
* Location of crest of free gingival margin in respect to CEJ.(REC) All clinical parameters were recorded at six sites (mesio-buccal, mid-buccal, disto-buccal, disto-lingual, mid-lingual and mesio-lingual) per tooth in all teeth except for third molars. BOP was assessed as a dichotomous measure (bleeding present or absent) within 15 seconds of probing. PD was recorded from gingival margin to base of pocket and CAL from cementoenamel junction (CEJ) to base of pocket.

PRIMARY AND SECONDARY OUTCOME VARIABLES Improvement in PPD and CAL over 6 months was considered as the primary outcome variable of the study. Secondary variables included improvement in PI, GI, BOP and REC.

PHASE 1 THERAPY Phase 1 therapy included patient education, motivation and plaque control. Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler (EMS Piezon 250 ,Switzerland), hand scaler and curettes (Hu-Friedy) was completed . Patients were kept on maintenance therapy.

All clinical parameters were recorded in 48 eligible patients after 8 weeks of SRP. A custom made acrylic stent was fabricated to standardized the location and angulations of periodontal probe. The study procedure was explained to the patient in their own language. Written and verbal informed consent was obtained from each patient. Patients were randomly allocated to test group and control group by envelop method. 48 labelled papers, 24 papers with label 1 and 24 papers with label 2 were placed into an envelope. If the patient picked paper with label 1 he or she was assigned to control group, while picking paper with label 2 meant assignment into test group.

PERIODONTAL SURGICAL PROCEDURE Modified Widman flap surgery was performed in both groups. After administration of local anaesthesia, first incision which is an internal bevel incision, was made 0.5 mm away from the crest of gingival margin to crest of alveolar bone, 2nd intra-crevicular incision from base of periodontal pocket to crest of alveolar bone and 3rd incision /horizontal incision follow the contour of the alveolar crest and the inter-proximal septum to cut loose the collar of gingival tissues which has been separated from the buccal or lingual flap and the teeth. A mucoperiosteal flap was reflected including at least one tooth ahead and one tooth behind the tooth/teeth involved. Meticulous debridement and root planning was carried out using area specific curettes and scalers to remove all the granulation tissue. After instrumentation, the root surface were washed with saline solution in attempt to remove any remaining detached fragments from the surgical field. After debridement mucoperiosteal flaps were repositioned and secured by using 3-0 non absorbable black silk surgical suture. Test group was given modified vertical internal mattress suture. The needle was passed through the buccal flap from the external surface, across the interdental area and through the lingual flap from the internal surface. The suture was run back to the buccal side by passing the needle through the lingual and buccal flaps .Thereafter, the suture is brought through the approximal site coronally to the tissue, passed through the loop of the suture on the lingual aspect, and then brought back to the starting point on the buccal side and tied. The control group was given simple loop interrupted interdental suture. The needle is passed through the buccal flap from the external surface, across the interdental area and the lingual flap from the internal surface or vice versa and tied. Post operative instructions were given.

Follow up was done after 3 and 6 months post-operatively.

STATISTICAL ANALYSIS :

All statistical analysis were carried out using statistical software (SPSS,Version 25.0 for Windows,SPSS,Chicago,IL).The normality of distribution of the data was assessed using the Shapiro-Wilk test. Data for PI, GI, BOP, PPD, CAL and REC followed non-normal distribution. Non-parametric tests were applied for PI, GI, PPD, CAL and REC. Wilcoxon-Signed Ranks test was applied for intragroup comparison and Mann Whitney test for intergroup comparison. Statistical analysis of BOP was done by McNemar test in intragroup and Chi-square test for intergroup comparison. Correlation and association between predictors and dependent variables was analysed by using Mixed Model analysis. Statistical significance level was set at P=0.05.

ELIGIBILITY:
Inclusion Criteria:.

* Systemically healthy individual possessing ≥20 natural teeth.
* Chronic periodontitis criteria as defined by division of Oral health at the centre for Disease Control and Prevention (CDC) in collaboration with American Academy of Periodontology (AAP) 42 (Page and Eke 2012) i.e.at least two or more interproximal sites with clinical attachment loss(CAL)≥4 mm (not on the same tooth),or ≥2 interproximal sites with probing pocket depth (PD)≥5 mm (not on the same
* Residual pocket depth ≥4 mm after phase 1 therapy for surgical intervention.

Exclusion Criteria:

* Patients with vertical bone loss.
* Current or former smokers or use of tobacco in any form.
* Patient on anti-inflammatory drugs or antibiotics or history of treatment with medication known to influence periodontal status or healing such as statins, glucocorticoids, phenytoin, calcium channel blockers, immunosuppressants, bisphosphonates or any other host modulatory drug within six months of commencement of study.
* Pregnant women, lactating mothers and women taking oral contraceptives.
* Patient who had undergone periodontal treatment within 6 months prior to the study.
* Patient with average plaque index ≥1.5 after phase 1 therapy.
* Miller Grade II /III tooth mobility after phase 1 treatment.
* Periapical infection in any tooth of the surgical treatment segment.

Ages: 30 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 6 months
  CAL was recorded from cementoenamel junction to base of pocket.

SECONDARY OUTCOMES:
Bleeding on probing | 6 months
  BOP was assessed as a dichotomous measure (bleeding present or absent) within 15 seconds of probing.

CONTACTS AND LOCATIONS:
Overall Officials: Krishan Kumar, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCE,ROHTAK,HARYANA,INDIA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India